CLINICAL TRIAL: NCT05512611
Title: Photopletysmography Detects Early Acute Blood Loss in Compensated Blood Donor Volunteers
Brief Title: Photoplethysmography for Diagnose Incipient Hypovolemia
Status: Completed | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: 2919-2809/2022
Record Dates: First submitted 2022-04-12; First posted 2022-08-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-03

CONDITIONS: Hypovolemia
Keywords: Photoplethysmography; Vital signs; Hemodynamics
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Finger photoplethysmography — Finger photoplethysmography in tested hand, noninvasive blood pressure and heart rate during blood donation.

SUMMARY:
Hypovolemia caused by acute bleeding increased morbi-mortality in emergency and operatin rooms. Precise real-time diagnosis of incipient acute hypovolemia is lacking at the bedside. We hypothesize that the infrared-red signals of pulse oximetry are sensitive to acute changes in patient's volemia. We aimed to test this hypothesis in a cohort of healthy blood donors as a model of simulated acute hypovolemia.

DETAILED DESCRIPTION:
This is a prospective and observational study designed to determine if the changes observed in finger photoplethysmographic waveform can detect incipient hypovolemia. The investigators will studied 60 blood donor volunteers as a model of slight hypovolemia (8-10% of the volemia). Vital signs and photoplethysmography will be recorded in the thumb of the tested hand during a standard blood donation protocol. Recorded data will be analyzed and compared before and after blood donation .

ELIGIBILITY:
Inclusion Criteria:

* Written Inform Consent
* weight > 50 kg,
* hemoglobin >12.5 gr/dl

Exclusion Criteria:

* pregnancy,
* ≤ 12 months from delivery or abortion,
* symptoms of allergy,
* fever >37 °C,
* infectious diseases,
* addictions,
* volunteers that received previous blood transfusions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy blood donor volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Analysis of the continuous component (DC) of the photoplethysmography signal. | 15 minutes
  The DC components of photoplethysmography is measured in arbitrary units (a.u).

SECONDARY OUTCOMES:
Analysis of non-invasive arterial blood pressure (NIBP) | 15 minutes
  NIBP is recorded in mmHg. This information is analyzed before and after blood donation.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Tusman, MD, Study Chair — Hospital Privado de Comunidad
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No